CLINICAL TRIAL: NCT02381522
Title: Remote Ischemic Pre-conditioning in Subarachnoid Hemorrhage
Acronym: RIPC-SAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Ronak Raval, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 5150015
Record Dates: First submitted 2015-02-13; First posted 2015-03-06 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Brain Aneurysms
Keywords: remote ischemic preconditioning
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Pre-conditioning (Active Comparator): Remote Ischemic Pre-conditioning group will receive 4 cycles of lower extremity occlusion of perfusion by blood pressure cuff inflated to 20 mmHg higher than systolic and confirmed by doppler.
  Interventions: Other: Remote Ischemic Pre-conditioning
- Sham RIPC (Sham Comparator): Sham procedure group will receive 4 cycles of inflation of lower extremity blood pressure cuff but it will be 20mmhg lower than systolic BP and hence not occlude the vessel.
  Interventions: Other: Sham RIPC

INTERVENTIONS:
Other: Remote Ischemic Pre-conditioning
  Arms: Remote Ischemic Pre-conditioning
Other: Sham RIPC
  Arms: Sham RIPC

SUMMARY:
The purpose of the study is to investigate if briefly stopping blood flow to the patient's leg will lead to the patient's body being better able to tolerate possible decreased blood flow to regions of the brain which otherwise frequently happens after subarachnoid hemorrhage.

Previous studies show that various organs such as the heart, brain or kidney can tolerate longer periods of decreased blood flow if prior to that insult shorter periods of decreased blood flow were experienced.

DETAILED DESCRIPTION:
Rupture of brain aneurysms is a common cause of death and disability, accounting for as many as 10% of stroke cases in the United States. While much of the resulting injury to the nervous system is caused by the initial bleeding from the aneurysm, many of these patients develop cerebral vasospasm, pathological constriction of the blood vessels supplying the brain, several days following hemorrhage. As many as a third of patients can suffer a resulting neurological deficit and stroke, presumably caused by the decreased blood flow to the brain (ischemia). This delayed brain injury accounts for a significant percentage of poor outcomes following aneurysm rupture. Remote ischemic preconditioning by transient limb ischemia (produced by inflation of a blood pressure cuff on the arm or leg) has been shown to minimize ischemic injury to other organs, most notably the heart. This "remote ischemic preconditioning" has the promise of protecting the brain from ischemic injury. Whereas in other forms of stroke the onset of ischemia cannot be predicted in the general population, following aneurysm rupture the investigators know patient's risk of developing vasospasm. Therefore, ischemic preconditioning following aneurysm rupture may help prevent some of the ischemic injury caused by vasospasm. One small study has shown decrease in vasospasm and metabolic products of ischemia in patients treated with remote ischemic preconditioning after subarachnoid hemorrhage. Decreased vasospasm due to remote ischemic preconditioning of the brain following aneurysm rupture still needs to be validated and question remains if that shows a mortality and morbidity benefit.

Remote Ischemic Preconditioning (RIPC) Procedure: Following enrollment, computer generated randomization will be done to see if the patient gets RIPC or sham-RIPC procedure. Patients will receive four cycles of lower limb remote ischemic preconditioning, starting at the earliest post-hemorrhage day. The remote ischemic preconditioning will typically take place on post-hemorrhage day 2 - 12. Each cycle of RIPC will consist of four 5-minute cycles of lower limb ischemia followed by 5-minute periods of reperfusion. A large manual bedside blood pressure cuff will be wrapped around the upper thigh of one leg. The cuff will be inflated to a pressure 20 mm Hg greater than the systolic arterial blood pressure measured by the patient's arterial line or upper limb blood pressure cuff. The adequate level of inflation will be confirmed by the absence of pulse in the ipsilateral pedal artery as detected by Doppler. The cuff will remain inflated for 5 minutes. The cuff will then be deflated and the limb will be allowed to re-perfuse for at least 5 minutes. After the cuff is deflated, the same procedure will then be repeated three times for a total of four cycles. Patients receiving the sham-RIPC procedure will have the cuff inflated to a pressure of 20 mmHg lower than systolic, hence to not occlude blood flow or cause ischemia. The rest of the study will be conducted similarly in both groups. Research staff will be aware if the patient is in the sham or treatment group. Patient, their nurse, treating physicians, lab technicians and Transcranial Doppler (TCD) technicians will not be made aware if the patient is receiving sham or treatment procedure.

Evaluation of Tolerance to the RIPC Maneuvers: The patient will be continuously monitored for pain and discomfort during the RIPC session. If the patient pain is more than 6 in the traditional 1-10 scale or if the patient expresses their desire to stop the maneuver, the procedure will be stopped, and the data regarding number and duration of the maneuvers will be recorded. A down-escalation of the treatment will be proposed, by reducing the number of cuff inflations to 3 or 2, as tolerated.

Hemodynamic evaluation of the effect of RIPC Maneuvers: Intracranial pressure (if bolt or external ventricular vein (EVD) present), blood pressure, oxygen saturation and heart rate will be monitored through the pre-conditioning process. If heart rate or BP changes greater than 20% of baseline and cannot be attributed to anything else the preconditioning will be stopped and allowed to normalize before retrying or be aborted based on bedside nurse, physicians, or research staff discretion. Oxygen saturation will also need to be above 92% at all times and ICP<20 when starting or at discretion of the bedside nurse or physician. Glascow Coma Score (GSC) will be monitored by nursing staff and recorded per ICU protocol. (TCD) measurements will be performed per ICU protocol.

Clinical assessments of the patients will be performed daily and at discharge from the ICU as per protocol. Modified Rankin Scale will be performed by research staff on arrival, Day 14, discharge, and by telephone at 1 and 6 months.

Data gathered from patients' chart will include location of aneurysm, interventions performed, Hunt & Hess score, Fisher grade determined by CT-head, PT/PTT/INR, chemistries and CBC (standard of care labs). Also information regarding ICU length of stay, hospital length of stay, Transcranial Doppler measurements, GCS during stay, mortality and demographics data will be gathered (includes age, sex, race, prior to admission Rankin score).

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Diagnosis of recent aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

1. Patients with a known history of lower limb vascular disease, lower limb vascular bypass surgery and/or peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Remote Ischemic Pre-Conditioning's effect on cerebral vasospasm as measured by Transcrananial Doppler (TCD) velocities. | 2 years
  RIPC or Sham RIPC will be done for two weeks or duration of patients hospital stay if shorter than 2 weeks. TCD measurements will be done during that time.

SECONDARY OUTCOMES:
Remote Ischemic Pre-conditioning's effect on functional outcome measured by Rankin Score | 2 years
  Rankin score will be assessed at 2 weeks, and by phone at one and six months.
Remote Ischemic Pre-conditioning's effect on complete blood count (CBC) | 2 years
  RIPC or Sham RIPC will be done for two weeks or duration of patients hospital stay if shorter than 2 weeks. CBC measurements will be done during that time.
Remote Ischemic Pre-conditioning's effect on basic metabolic panel (BMP) | 2 years
  RIPC or Sham RIPC will be done for two weeks or duration of patients hospital stay if shorter than 2 weeks. BMP measurements will be done during that time.
Remote Ischemic Pre-conditioning's effect on coagulation parameters | 2 years
  RIPC or Sham RIPC will be done for two weeks or duration of patients hospital stay if shorter than 2 weeks. Coagulation parameter measurements will be done during that time.
Remote Ischemic Pre-conditioning's effect on GCS | 2 years
  RIPC or Sham RIPC will be done for two weeks or duration of patients hospital stay if shorter than 2 weeks. GCS measurements will be done per ICU protocol during that time and they will be recorded.
Remote Ischemic Pre-conditioning's effect on mortality | 2 years
  Total six months of follow up will be done and this will be the time mortality is assessed.
Remote Ischemic Pre-conditioning's effect on needing additional angiographic intervention | 2 years
  RIPC or Sham RIPC will be done for two weeks or duration of patients hospital stay if shorter than 2 weeks. Need for additional angiographic intervention during this period will be recorded.
Remote Ischemic Pre-conditioning's effect on additional neurological events | 2 years
  Total six months of follow up will be done and additional neurological events during this time period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Raval, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States